CLINICAL TRIAL: NCT00090675
Title: A Phase IIIb Randomized, Double-Blind Study Comparing Maintenance ZD1839 (IRESSA®) or Placebo Following Completion of Front Line, Platinum-Based, Double Chemotherapy in Subjects With Advanced or Metastatic Non-Small Cell Lung Cancer
Brief Title: Maintenance ZD1839 (IRESSA®) Following Completion of Front Line, Platinum-Based, Double Chemotherapy in Subjects With Advanced or Metastatic Non-Small Cell Lung Cancer
Acronym: IMAC/Herbst
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: No patients randomised
Sponsor: AstraZeneca (Industry)
Allocation: Randomized | Masking: Double | Purpose: Treatment
Other Study IDs: D7913L00019; Herbst trial
Record Dates: First submitted 2004-09-02; First posted 2004-09-03 (Estimated); Last update posted 2013-01-29 (Estimated); Status verified 2013-01

CONDITIONS: Non-Small-Cell Lung Carcinoma
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Gefitinib

INTERVENTIONS:
Drug: ZD1839

SUMMARY:
In this Phase IIIb, randomized, double-blind, maintenance study, 300 subjects with advanced or metastatic Non-Small Cell Lung Cancer (NSCLC) (Stage IIIB {T4-pleural effusion} and IV) who have SD or objective tumor response immediately following the completion of 4-6 cycles of front line, platinum-based, doublet chemotherapy will be randomized in a double-blind manner to receive either ZD1839 or placebo.

ELIGIBILITY:
Inclusion Criteria:

* Must sign Informed Consent
* Females and males aged 18 years and over.
* Confirmed stage IIIB (T4-pleural effusion) and IV NSCLC.
* Either complete response, partial response, or stable disease following at least 4 cycles (3 in the setting of intolerable toxicity) but no more than 6 cycles of definitive front line, platinum-based, doublet chemotherapy.
* No prior EGFR therapy
* No newly diagnosed intracerebral metastases while receiving or after completing chemotherapy
* At least 3 weeks (21 days) but no more than 4 weeks (28 days) since last dose of chemotherapy
* Must be completely healed from previous major oncologic surgery
* Life expectancy of ≥ 8 weeks.

Exclusion Criteria:

* Known severe hypersensitivity to ZD1839 or any of the excipients of these products.
* Any evidence of clinically active interstitial lung disease (subjects with chronic, stable, radiographic changes who are asymptomatic need not be excluded).
* Other co-existing malignancies or malignancies diagnosed within the last 5 years with the exception of basal cell carcinoma or cervical cancer in situ.
* Any unresolved chronic toxicity greater than common toxicity criteria (CTC) grade 2 from previous anticancer therapy excluding peripheral neuropathy or alopecia.
* Evidence of any significant clinical disorder or laboratory finding that makes it undesirable for the subject to participate in the study.
* Pregnancy or breast feeding (women of child bearing potential). Women of childbearing potential must practice acceptable methods of birth control to prevent pregnancy.
* Treatment with a non-approved or investigational drug within 30 days before Day 1 of study treatment.
* Signs of neurological symptoms consistent with new onset spinal cord compression or CNS metastases.
* Treatment with any systemic anticancer therapies other than the prescribed protocol chemotherapy regimen (refer to Inclusion criterion -). Exception: Palliative radiotherapy for symptom relief of lesions present at diagnosis will be allowed; however, this radiotherapy must occur prior to completion of pre-study doublet chemotherapy.
* Males must also be willing to practice acceptable methods of birth control while taking the drug to prevent pregnancy of a partner.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2006-01; Primary Completion 2007-11 (Estimated); Study Completion 2007-11 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Iressa Medical Science Director, Study Director — AstraZeneca